CLINICAL TRIAL: NCT00306670
Title: A Prospective, Phase II/III Randomized, Mult-institutional Controlled, Open-label, Phase II Trial of Rituximab Versus Oral Cyclophosphamide to Eradicate or Suppress Autoimmune Anti-Factor VIII Antibodies in Patients With Acquired Hemophilia A
Brief Title: Trial of Rituximab Versus Oral Cyclophosphamide to Eradicate or Suppress Autoimmune Anti-Factor VIII Antibodies in Acquired Hemophilia A
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor no longer funding study.
Sponsor: Georgetown University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Craig Kessler, Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U2688
Record Dates: First submitted 2006-03-23; First posted 2006-03-24 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Hemophilia A
Keywords: Acquired Hemophilia A; Anti-Factor VIII antibodies; Anti-Factor VIII inhibitors; Hemophilia A; Factor VIII inhibitors
MeSH Terms: conditions — Hemophilia A; Factor 8 deficiency, acquired | interventions — Rituximab; Prednisone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rituximab (Experimental): Patients will receive rituximab.
  Interventions: Drug: Rituxan; Drug: prednisone
- Oral cyclophosphamide (Active Comparator): Patients will receive oral cyclophosphamide.
  Interventions: Drug: prednisone

INTERVENTIONS:
Drug: Rituxan — Acquired Hemophilia A Patients Who Have Developed Anti-Factor VIII Antibodies
  Other Names: Rituximab
  Arms: Rituximab
Drug: prednisone — <30 mg/day
  Other Names: corticosteroids

SUMMARY:
The purpose of this study is to evaluate the rate of response when administering rituximab to suppress or eliminate the anti-body in a patient's blood that inhibits the effectiveness of their factor replacement product compared to treatment using cyclophosphamide. This is a Phase 2/3 study to find out what effects (good and bad) and response rituximab has on a patient and their anti-Factor VIII antibodies. Also, to compare the effect (good and bad) of the rituximab with cyclophosphamide on a patient and their anti-Factor VIII antibodies to see which is better. This research is being done because we do not know which treatment regimen (rituximab or cyclophosphamide) is more effective in eliminating or suppressing the anti-Factor VIII antibody in patients with acquired Hemophilia A.

DETAILED DESCRIPTION:
This is a prospective Phase II randomized multi-institutional controlled pilot trial comparing the regimen of single agent rituximab with 6 weeks cytotoxic therapy with oral cyclophosphamide to eradicate or suppress autoimmune anti-factor VIII antibodies in individuals with acquired hemophilia A. Patients will be randomized to receive either of these two regimens when their autoimmune anti-factor VIII antibodies prove to be refractory to initial upfront immunosuppressive treatment with oral prednisone 1 mg/kg/day (or equivalent corticosteroid doses) for 3 weeks. Patients will be randomized to the treatment cohorts according to the biostatistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acquired hemophilia A in a previously non-coagulopathic individual.
* Prior treatment with at least 3 weeks of immunosuppressive therapy
* Factor VIII: C levels <50% within 14 days prior to study entry, which do not correct in coagulation assays in which normal plasma is mixed and incubated with patient plasma.
* Measurable anti-factor VIII:C antibody inhibitor activity > 0.6 Bethesda Units/ml.
* Age ³18 years
* Written informed consent
* Use of an effective means to avoid pregnancy, including abstinence, for women of childbearing potential,.
* Serum bilirubin less than or equal to the upper limit of normal (ULN); ALT and AST £2.5´ ULN within 14 days prior to study entry
* Serum creatinine £1.5´ the ULN within 14 days prior to study entry
* Negative serum pregnancy test, for all women of childbearing potential, within 14 days prior to study entry

Exclusion Criteria:

* Continued treatment requirement of prednisone ≥30mg/day or equivalent dosing of other corticosteroid preparations to control serious symptoms of an underlying autoimmune disease state.
* Treatment with cyclophosphamide, danazol, vinca alkaloids, azathioprine, IVIG, or other immunosuppressive, immunomodulatory, or cytotoxic agents (other than decreasing doses of corticosteroids) within 30 days prior to study entry.
* Anticipated need for repeated extracorporeal plasmapheresis in order to reverse refractory bleeding associated with acquired hemophilia.
* Treatment with other experimental agents within 30 days prior to study entry
* Known sensitivity to murine or chimeric products
* Hepatitis BsAg positivity or high risk for reactivation of Hepatitis B.
* Active infection requiring antibiotic therapy within 7 days prior to study entry
* Current use of any required medications, which in the opinion of the treating physician, could be inducing the formation of auto-FVIII:C inhibitory antibodies
* Prior treatment with rituximab or other monoclonal antibody therapy
* Known HIV antibody positivity
* NCI-CTC Grade ³1 cardiac arrhythmia ( refer to CTC v3)
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Currently pregnant women, lactating women, or women within 12 months of delivery, spontaneous miscarriage, or therapeutic or elective termination of pregnancy.
* Known severe leucopenia (absolute neutrophil count <1000/µL) or thrombocytopenia (<25,000/µL);
* Known pre-existing cystitis or severe urinary outflow obstruction.
* Known history of recurrent severe opportunistic infections, eg. generalized herpes zoster;
* Inability or unwillingness to comply with study design and requirements and follow-up procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-04; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Kessler, MD, Principal Investigator — Georgetown University Hospital

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab | Oral Cyclophosphamide
Started | 0 (no patients recruited; Genentech, the study sponsor, pulled funding and discontinued the protocol) | 2 (2 patients recruited; Genentech, the study sponsor, discontinued trial before treatment started)
Completed | 0 (no patients recruited; Genentech, the study sponsor, pulled funding and discontinued the protocol) | 0 (2 patients recruited; Genentech, the study sponsor, discontinued study before treatment initiated)
Not Completed | 0 | 2
Not completed — patients recruited; Genentech, the st | 0 | 2

BASELINE CHARACTERISTICS:
Population: Patients diagnosed with acquired FVIII inhibitors were to be randomized to Rituximab versus oral cyclophosphamide to evaluate efficacy of inhibitor eradication and safety
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | Oral Cyclophosphamide | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Continuous [Mean (Full Range); unit: years] |  | 60 [52 to 68] | 60 [52 to 68]
Gender [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 2 | 2
factor VIII activity; factor VIII inhibitor titer [Mean (Full Range); unit: units on a scale] |  | 25 [5 to 30] | 25 [5 to 30]

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Total Number of Circulating Lymphocytes and Lymphocyte Phenotypes and to Correlate With the Effectiveness of Rituximab and Oral Cyclophosphamide to Achieve and Preserve Complete Eradication of the Refractory Autoantibody.
Description: the 2 recruited patients did not eradicate their inhibitors with 3 weeks of corticosteroids and did not progress in clinical trial since funding was eliminated and study terminated
Time Frame: When 25 patients have completed the study.
Population: 2 patients with acquired hemophilia A: two patients were recruited, but the sponsor terminated the study before the patients started treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Oral Cyclophosphamide
Number analyzed (Participants) | 0 | 2
Participants |  | 0

ADVERSE EVENTS:
Arm/Group | Rituximab | Oral Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Sponsor terminated study prior to patient receiving first dose of study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No